CLINICAL TRIAL: NCT00790608
Title: A Phase II Trial on the Reduction of Methicillin Resistant Staphylococcus Aureus in MRSA Positive Ulcers
Brief Title: Clinical Trial on the Reduction of Methicillin Resistant Staphylococcus Aureus (MRSA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited recruitment
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP 5; EudraCT 2008-001287-36
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Skin Ulcers; Methicillin-resistant Staphylococcus Aureus Infection
MeSH Terms: conditions — Skin Ulcer | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nitric Oxide — Gaseous nitric oxide (1%), delivered for 30 minutes per day for 3 consecutive days

SUMMARY:
The purpose of the study is to determine if topically applied nitric oxide gas is effective in reducing the quantity of bacteria (including MRSA)in a wound.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent
* Must be ≥ 18 years of age and not of child bearing potential
* Must have an ulcer in which the presence of MRSA has been identified, but which is not clinically infected
* Must have an ulcer size not to extend beyond the inner borders of the dressing

Exclusion Criteria:

* Is a female of child bearing years or who could become pregnant
* Is < 18 years of age
* Has an clinically infected skin ulcer
* Has a ulcer that is being treated with a topical antimicrobial agent or has been treated with a topical antimicrobial agent during 3 days prior to enrolment
* Has been using systemic antibiotics during 7 days prior to enrolment into this study
* Has an ulcer which is identified as malignant in origin (e.g. Marjolin's ulcer)
* Has an ulcer size beyond the inner borders of the dressing
* Is septic or has other signs of an invasive infection
* Has used any investigational drug within 30 days preceding study participation.
* Suffers from a condition, which, in the opinion of the Investigator, would compromise his or her safety.
* Suffers from a condition which, in the opinion of the Investigator, would compromise the quality of the data.
* Has a known allergy to any of the products that are part of this protocol
* Suffers from a condition which, in the opinion of the Investigator, would seriously interfere negatively with the normal parameters of immune response to an infection.
* Is using any of the prohibited concomitant medications or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in bioburden (specifically MRSA)as assessed via quantitative cultures. | 10 Days

SECONDARY OUTCOMES:
Improvement in the condition of the ulcer as judged by comparative photography and independent clinical assessment | 10 Days
Incidence of adverse events | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, MB ChB, MRGCP, FRCS, Principal Investigator — Department of Wound Healing, Cardiff University
Locations (1):
- Department of Wound Healing, Cardiff University, Cardiff, United Kingdom